CLINICAL TRIAL: NCT02479061
Title: An Observational Study of the Prevalence of Patients Requiring Palliative Care in the French Anti Cancer Centers.
Brief Title: An Observational Study of the Prevalence of Patients Requiring Palliative Care in French Anti-cancer Centers.
Acronym: PREPA-10
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: PREPA-10
Record Dates: First submitted 2015-06-19; First posted 2015-06-23 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Neoplasms; Oncology
Keywords: Observationnal study; Prevalence; Palliative care; Anti cancer center
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to determine the proportion of patients with a score greater than 3/10 to the questionnaire PALLIA-10.

This questionnaire is a tool provided by the French Society for Palliative Cares, aiming at helping the providers of care to identify patients who would require palliative cares.

According to the notice of the questionnaire, patients with a score greater than 3 would be taken in charge by a palliative care team. Considerong the 10 itmes of this questionnaire, it seems that a large majority of patients would have a score greater than 3 in the context of anti cancer centers.

To date, palliative teams are not designed to take in charge such an amount of patients.

DETAILED DESCRIPTION:
Continuous improvement of therapeutics helped to lengthen different stages of natural cancer evolution. Advanced cancer patients are followed-up even longer; therefore there is a need to increase palliative care resources. A global therapeutic approach is being set up gradually thanks to specialized supportive care team. This global approach includes therapeutics and life condition improvement of the patient and his family.

In France, only 2 anti-cancer centers have a palliative care unit. The 16 other centers design hospital beds for palliative care and work with mobile palliative care teams.

According to latest studies with high level of evidence, International oncology societies published good practices guidelines supporting the need of early palliative cares for patients with metastatic cancer.

In 2010, Temel et al. demonstrated early palliative care effectiveness. Indeed, early palliative care led to significant improvements in both quality of life (score on the FACT-L scale: 98.0 vs. 91.5; p=0.03) and mood (depressive symptoms: 16% vs. 38%, P=0.01). Moreover median survival was longer among patients receiving early palliative care (11.6 months vs. 8.9 months, p=0.02). Analysis showed that patients assigned to early palliative care stopped chemotherapy earlier, had a higher enrollment rate in palliative care units and less depressive symptoms when cares were provided by both oncologists and palliative care teams.

Other specific scales support efficiency of early palliative care on quality of life. Early palliative care increases also satisfaction of the cares. Therefore, these results illustrate the need for an early integration of palliative care in France; and this approach is recommended in the third national plan against cancer.

Despite efficacy data, no high international consensus exists on a screening score for patients requiring early palliative care. Some teams therefore use prognostic factors like Barbot score.

Confronted with such difficulties, the French Society for Counselling and Palliative Care create a score (PALLIA-10) with 10 items on personal situation of the patient and his disease. This score helps medical staffs to direct patients to a specialized team as soon as it is > 3/10.

PALLI-10 score is not optimized because of the large number of patients with a score > 3 in the French anti-cancer centers. In 2014, a team from Centre Fraçois Baclesse (Caen, France) showed that nearly 65% of hospitalized patients in medicine department has a score PALLIA-10 > 3/10. Today, mobile palliative care teams are too small to manage so many patients.

First, it is important to evaluate the prevalence of these patients in France. Description of patients hospitalized in a Center for the Treatment of Cancers should help us to describe the characteristics of patients requiring cares provided by a mobile palliative care team.

ELIGIBILITY:
Inclusion Criteria:

* 18-year old or older
* Hospitalized in a conventionnal medical service, including radiotherapy, brachytherapy, palliative care units.

Exclusion Criteria:

* Patient hospitalized in an out-patient service, surgery unit, weekly units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized in a conventionnal medical service of a French anti cancer center.
Sampling Method: Non-Probability Sample
Enrollment: 846 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a score greater than 3/10 to questionnaire PALLIA-10 in the population of patients hospitalized in a French cancer center. | Day 1 of the study

SECONDARY OUTCOMES:
The proportion of patients with a score greater than 5 to questionnaire PALLIA-10 | Day 1 of the study
Proportion of patients already followed-up by a palliative care team | Day 1 of the study
Mean score to questionnaire PALLIA-10 | Day 1 of the study
Predictive factors of current palliative cares | Day 1 of the study
Prognostic factors of overall survival | From Day 1 of the study to the update of survival status (6 months later)

CONTACTS AND LOCATIONS:
Overall Officials: Gisele CHVETZOFF, MD, Principal Investigator — Centre Leon Berard
Locations (15):
- France (15):
  - Institut de Cancérologie de l'Ouest, Angers
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean PERRIN, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris - Saint Cloud
  - Institut Jean GODINOT, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Paul Strauss, Strasbourg
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No